CLINICAL TRIAL: NCT03255967
Title: A Multisite Cluster RCT of the Dementia Symptom Management at Home Program
Brief Title: Dementia Symptom Management at Home Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 17-00810
Record Dates: First submitted 2017-08-15; First posted 2017-08-21 (Actual); Results first posted 2024-01-30 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Dementia
MeSH Terms: conditions — Dementia | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- QI program care (Experimental): DSM-H performance improvement program Patients in the performance improvement group will receive care from a care team who has received the DSM-H performance improvement program
  Interventions: Behavioral: DSM-H
- Control (Active Comparator): Receive usual care from a care team who has not received the performance improvement program
  Interventions: Behavioral: Standard of Care

INTERVENTIONS:
Behavioral: DSM-H — Multi-modal quality improvement program for improving the quality of care provided to person with dementia (PWD)-informal caregiver dyads through HHC
  Arms: QI program care
Behavioral: Standard of Care — Subjects receive care through usual home healthcare assignment process.
  Arms: Control

SUMMARY:
Alzheimer's Disease and Related Disorders (dementia) poses a significant challenge to our public health. While many persons with dementia are cared for by friends and family in the community with the assistance of home healthcare, most home healthcare clinicians and agencies are ill prepared to care for this population and therefore have difficulty assisting patients and caregivers in maintaining quality of life leading to adverse patient outcomes, increased caregiver stress and burnout, and healthcare utilization. This study will therefore utilize a cluster randomized controlled design at 3 study sites to examine the ability of a multi-component evidence-based practice primary palliative care quality improvement program for home healthcare registered nurses, occupational therapists and physical therapists to improve the quality of life and reduce healthcare utilization for persons with dementia and their informal caregiver.

ELIGIBILITY:
Inclusion Criteria:

* PWD over the age of 65
* Admitted to one of the three HHC agencies
* The patient and family caregiver speak English and/or Spanish.
* The informal caregiver is ≥18 years of age and spends at least 8 hours per week with the patient.
* Patients who score ≥6 on the Quick Dementia Rating Scale (at least mild impairment).

Exclusion Criteria:

* Patients with a separate Axis 1 diagnosis other than forms of dementia, depression or anxiety.
* PWD residing in assisted living facilities or board and care homes
* PWD solely receiving infusion or home health aide services.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 217 (Actual)
Dates: Start 2018-08-16 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Abraham Brody, MD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States

REFERENCES:
- [Derived] Bristol AA, Convery KA, Sotelo V, Schneider CE, Lin SY, Fletcher J, Rupper R, Galvin JE, Brody AA. Protocol for an embedded pragmatic clinical trial to test the effectiveness of Aliviado Dementia Care in improving quality of life for persons living with dementia and their informal caregivers. Contemp Clin Trials. 2020 Jun;93:106005. doi: 10.1016/j.cct.2020.106005. Epub 2020 Apr 19. PMID 32320844

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The trial enrolled 215 Patient-Caregiver Dyads (215 patients with dementia (PWD) and 215 caregivers). 119 Dyads were randomized to the QI program care arm and 96 Dyads were randomized to the Control arm.
Groups:
- QI Program Care: DSM-H performance improvement program Patients in the performance improvement group will receive care from a care team who has received the DSM-H performance improvement program
  DSM-H: Multi-modal quality improvement program for improving the quality of care provided to PWD-informal caregiver dyads through HHC
Period: Overall Study
Arm/Group | QI Program Care | Control
Started | 238 | 192
Number of Patients Started | 119 | 96
Number of Patients Completed | 99 | 76
Number of Caregivers Started | 119 | 96
Number of Caregivers Completed | 99 | 76
Completed | 198 | 152
Not Completed | 40 | 40
Not completed — Adverse Event | 26 | 30
Not completed — Withdrawal by Subject | 6 | 6
Not completed — Schedule conflict | 6 | 4
Not completed — POA did not sign consent form | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- QI Program Care - PWD: Patients with dementia (PWD) assigned to the QI program care arm as part of a Patient-Caregiver dyad.
- QI Program Care - Caregiver: Caregivers assigned to the QI program care arm as part of a Patient-Caregiver dyad.
- Control - PWD: Patients with dementia (PWD) assigned to the control arm as part of a Patient-Caregiver dyad.
- Control - Caregiver: Caregivers assigned to the control arm as part of a Patient-Caregiver dyad.
- Total: Total of all reporting groups
Arm/Group | QI Program Care - PWD | QI Program Care - Caregiver | Control - PWD | Control - Caregiver | Total
Number analyzed (Participants) | 119 | 119 | 96 | 96 | 430
Age, Continuous [Mean (Standard Deviation); unit: years] | 83 (7.3) | 63 (13.7) | 84 (7.9) | 57 (11.9) | 71.75 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 74 | 92 | 63 | 73 | 302
  Male | 45 | 27 | 33 | 23 | 128
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 16 | 15 | 12 | 12 | 55
  Not Hispanic or Latino | 103 | 104 | 84 | 84 | 375
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 2 | 2 | 2 | 2 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 35 | 35 | 27 | 27 | 124
  White | 74 | 73 | 62 | 62 | 271
  More than one race | 2 | 2 | 2 | 2 | 8
  Unknown or Not Reported | 6 | 7 | 3 | 3 | 19
Region of Enrollment [Number; unit: participants]
  United States | 119 | 119 | 96 | 96 | 430

OUTCOME MEASURES:

1. Primary Outcome: Change in Quality of Life-Alzheimer's Disease Score
Description: 13-item measurement of Alzheimer's disease patients' health-related quality of life (HRQOL) by proxy (caregiver) assessment. Each item is rated on a 4-point Likert scale ranging from 1 (poor) to 4 (excellent). The total score is the sum of responses and ranges from 13 to 52; higher scores indicate greater HRQOL. An increase in scores indicates HRQOL increased during the observational period.
Time Frame: Baseline, Day 60
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | QI Program Care | Control
Number analyzed (Participants) | 119 | 96
score on a scale | 12.32 (16.69) | 15.88 (22.77)

2. Primary Outcome: Change in Caregiver-Targeted Quality of Life Measure Score - IADL Scale
Description: The Caregiver-Targeted Quality of Life (CG-QOL) measure covers 10 dimensions of QOL relevant to caregivers of persons with dementia. The CG-QOL comprises 80 items distributed across the following scales: assistance with activities of daily living (ADLs), assistance with instrumental ADLs (IADLs), personal time, role limitation due to caregiving, family involvement, demands of caregiving, worry, caregiver feelings, spirituality and faith, benefits of caregiving. The total score for the IADL scale ranges from 0-100; higher scores indicate greater quality of life. An increase in scores indicates quality of life with respect to assistance with IADLs improved during the observational period.
Time Frame: Baseline, Day 60
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | QI Program Care | Control
Number analyzed (Participants) | 119 | 96
score on a scale | 12.32 (16.69) | 15.88 (22.77)

3. Primary Outcome: Change in Caregiver-Targeted Quality of Life Measure Score - ADL Scale
Description: The Caregiver-Targeted Quality of Life (CG-QOL) measure covers 10 dimensions of QOL relevant to caregivers of persons with dementia. The CG-QOL comprises 80 items distributed across the following scales: assistance with activities of daily living (ADLs), assistance with instrumental ADLs (IADLs), personal time, role limitation due to caregiving, family involvement, demands of caregiving, worry, caregiver feelings, spirituality and faith, benefits of caregiving. The total score for the ADL scale ranges from 0-100; higher scores indicate greater quality of life. An increase in scores indicates quality of life with respect to assistance with ADLs improved during the observational period.
Time Frame: Baseline, Day 60
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | QI Program Care | Control
Number analyzed (Participants) | 119 | 96
score on a scale | 47.45 (37.45) | 44.94 (37.26)

4. Primary Outcome: Change in Caregiver-Targeted Quality of Life Measure Score - Role Limitations Scale
Description: The Caregiver-Targeted Quality of Life (CG-QOL) measure covers 10 dimensions of QOL relevant to caregivers of persons with dementia. The CG-QOL comprises 80 items distributed across the following scales: assistance with activities of daily living (ADLs), assistance with instrumental ADLs (IADLs), personal time, role limitation due to caregiving, family involvement, demands of caregiving, worry, caregiver feelings, spirituality and faith, benefits of caregiving. The total score for the role limitations scale ranges from 0-100; higher scores indicate greater quality of life. An increase in scores indicates quality of life with respect to role limitation due to caregiving improved during the observational period.
Time Frame: Baseline, Day 60
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | QI Program Care | Control
Number analyzed (Participants) | 119 | 96
score on a scale | 46.33 (28.96) | 46.56 (26.76)

5. Primary Outcome: Change in Caregiver-Targeted Quality of Life Measure Score - Personal Time Scale
Description: The Caregiver-Targeted Quality of Life (CG-QOL) measure covers 10 dimensions of QOL relevant to caregivers of persons with dementia. The CG-QOL comprises 80 items distributed across the following scales: assistance with activities of daily living (ADLs), assistance with instrumental ADLs (IADLs), personal time, role limitation due to caregiving, family involvement, demands of caregiving, worry, caregiver feelings, spirituality and faith, benefits of caregiving. The total score for the personal time scale ranges from 0-100; higher scores indicate greater quality of life. An increase in scores indicates quality of life with respect to personal care improved during the observational period.
Time Frame: Baseline, Day 60
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | QI Program Care | Control
Number analyzed (Participants) | 119 | 96
score on a scale | 38.71 (22.12) | 40.34 (19.67)

6. Primary Outcome: Change in Caregiver-Targeted Quality of Life Measure Score - Family Interaction Scale
Description: The Caregiver-Targeted Quality of Life (CG-QOL) measure covers 10 dimensions of QOL relevant to caregivers of persons with dementia. The CG-QOL comprises 80 items distributed across the following scales: assistance with activities of daily living (ADLs), assistance with instrumental ADLs (IADLs), personal time, role limitation due to caregiving, family involvement, demands of caregiving, worry, caregiver feelings, spirituality and faith, benefits of caregiving. The total score for the family interaction scale ranges from 0-100; higher scores indicate greater quality of life. An increase in scores indicates quality of life with respect to family interaction improved during the observational period.
Time Frame: Baseline, Day 60
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | QI Program Care | Control
Number analyzed (Participants) | 119 | 96
score on a scale | 53.27 (28.45) | 52.11 (28.42)

7. Primary Outcome: Change in Caregiver-Targeted Quality of Life Measure Score - Demands of Caregiving Scale
Description: The Caregiver-Targeted Quality of Life (CG-QOL) measure covers 10 dimensions of QOL relevant to caregivers of persons with dementia. The CG-QOL comprises 80 items distributed across the following scales: assistance with activities of daily living (ADLs), assistance with instrumental ADLs (IADLs), personal time, role limitation due to caregiving, family involvement, demands of caregiving, worry, caregiver feelings, spirituality and faith, benefits of caregiving. The total score for the demands of caregiving scale ranges from 0-100; higher scores indicate greater quality of life. An increase in scores indicates quality of life with respect to demands of caregiving improved during the observational period.
Time Frame: Baseline, Day 60
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | QI Program Care | Control
Number analyzed (Participants) | 119 | 96
score on a scale | 56.6 (24.39) | 56.22 (25.35)

8. Primary Outcome: Change in Caregiver-Targeted Quality of Life Measure Score - Worry Scale
Description: The Caregiver-Targeted Quality of Life (CG-QOL) measure covers 10 dimensions of QOL relevant to caregivers of persons with dementia. The CG-QOL comprises 80 items distributed across the following scales: assistance with activities of daily living (ADLs), assistance with instrumental ADLs (IADLs), personal time, role limitation due to caregiving, family involvement, demands of caregiving, worry, caregiver feelings, spirituality and faith, benefits of caregiving. The total score for the worry scale ranges from 0-100; higher scores indicate greater quality of life. An increase in scores indicates quality of life with respect to worry improved during the observational period.
Time Frame: Baseline, Day 60
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | QI Program Care | Control
Number analyzed (Participants) | 119 | 96
score on a scale | 51.25 (21.7) | 52.56 (19.89)

9. Primary Outcome: Change in Caregiver-Targeted Quality of Life Measure Score - Spirituality Scale
Description: The Caregiver-Targeted Quality of Life (CG-QOL) measure covers 10 dimensions of QOL relevant to caregivers of persons with dementia. The CG-QOL comprises 80 items distributed across the following scales: assistance with activities of daily living (ADLs), assistance with instrumental ADLs (IADLs), personal time, role limitation due to caregiving, family involvement, demands of caregiving, worry, caregiver feelings, spirituality and faith, benefits of caregiving. The total score for the spirituality scale ranges from 0-100; higher scores indicate greater quality of life. An increase in scores indicates quality of life with respect to spirituality improved during the observational period.
Time Frame: Baseline, Day 60
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | QI Program Care | Control
Number analyzed (Participants) | 119 | 96
score on a scale | 79.25 (29.1) | 67.75 (33.94)

10. Primary Outcome: Change in Caregiver-Targeted Quality of Life Measure Score - Benefits of Caregiving Scale
Description: The Caregiver-Targeted Quality of Life (CG-QOL) measure covers 10 dimensions of QOL relevant to caregivers of persons with dementia. The CG-QOL comprises 80 items distributed across the following scales: assistance with activities of daily living (ADLs), assistance with instrumental ADLs (IADLs), personal time, role limitation due to caregiving, family involvement, demands of caregiving, worry, caregiver feelings, spirituality and faith, benefits of caregiving. The total score for the benefits of caregiving scale ranges from 0-100; higher scores indicate greater quality of life. An increase in scores indicates quality of life with respect to benefits of caregiving improved during the observational period.
Time Frame: Baseline, Day 60
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | QI Program Care | Control
Number analyzed (Participants) | 119 | 96
score on a scale | 81.38 (20.18) | 79.34 (20.64)

11. Primary Outcome: Change in Caregiver-Targeted Quality of Life Measure Score - Caregiver Feelings Scale
Description: The Caregiver-Targeted Quality of Life (CG-QOL) measure covers 10 dimensions of QOL relevant to caregivers of persons with dementia. The CG-QOL comprises 80 items distributed across the following scales: assistance with activities of daily living (ADLs), assistance with instrumental ADLs (IADLs), personal time, role limitation due to caregiving, family involvement, demands of caregiving, worry, caregiver feelings, spirituality and faith, benefits of caregiving. The total score for the caregiver feelings scale ranges from 0-100; higher scores indicate greater quality of life. An increase in scores indicates quality of life with respect to caregiver feelings improved during the observational period.
Time Frame: Baseline, Day 60
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | QI Program Care | Control
Number analyzed (Participants) | 119 | 96
score on a scale | 72.53 (16.82) | 76.49 (13.73)

12. Primary Outcome: Number of Emergency Room (ER) Visits by Patients With Dementia (PWD) During Study Period
Description: Measured through interviews with the informal caregiver using the Resource Utilization Inventory.
Time Frame: Up to Day 60
Measure: Mean (Standard Deviation); unit: ER visits
Arm/Group | QI Program Care | Control
Number analyzed (Participants) | 119 | 96
ER visits | 0.08 (0.34) | 0.08 (0.31)

13. Primary Outcome: Number of PWD Inpatient Admissions During Study Period
Description: Measured through interviews with the informal caregiver using the Resource Utilization Inventory.
Time Frame: Up to Day 60
Measure: Mean (Standard Deviation); unit: Hospitalizations
Arm/Group | QI Program Care | Control
Number analyzed (Participants) | 119 | 96
Hospitalizations | 0.08 (0.4) | 0.13 (0.38)

14. Secondary Outcome: Change in Pain Assessment In Advanced Dementia (PAINAD) Score
Description: 5-item assessment of pain in individuals with advanced dementia. Items are ranked on a 3-point Likert scale from 0 to 2. The total score is the sum of responses and ranges from 0 (no pain) to 10 (severe pain). An increase in scores indicates pain increased during the observational period.
Time Frame: Baseline, Day 60
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | QI Program Care | Control
Number analyzed (Participants) | 107 | 85
score on a scale | 0.14 (0.62) | 0.05 (0.28)

15. Secondary Outcome: Change in Neuropsychiatric Inventory Questionnaire (NPI-Q) Score
Description: 13-item tool that measures caregiver perceptions of Behavioral and Psychological Symptoms of Dementia (BPSD). For each item, The severity of the reported symptoms is assessed on a 3-point scale. The total severity score ranges from 0 to 36 with higher scores representing worse severity. An increase in score indicates severity of BPSD increased during the observational period.
Time Frame: Baseline, Day 60
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | QI Program Care | Control
Number analyzed (Participants) | 117 | 96
score on a scale | 8.45 (6.31) | 7.96 (5.78)

16. Secondary Outcome: Number of PWD Who Use Antipsychotics During Study Period
Description: Measured via patient medication record.
Time Frame: Up to Day 60
Measure: Count of Participants; unit: Participants
Arm/Group | QI Program Care | Control
Number analyzed (Participants) | 119 | 96
Participants | 20 | 11

17. Secondary Outcome: Number of PWD Who Use Analgesics During Study Period
Description: Measured via patient medication record.
Time Frame: Up to Day 60
Measure: Count of Participants; unit: Participants
Arm/Group | QI Program Care | Control
Number analyzed (Participants) | 119 | 96
Participants | 45 | 39

18. Secondary Outcome: Number of PWD Outpatient Visits During Study Period
Time Frame: Up to Day 60
Measure: Mean (Standard Deviation); unit: Outpatient Visits
Arm/Group | QI Program Care | Control
Number analyzed (Participants) | 119 | 96
Outpatient Visits | 4.5 (12.15) | 3.16 (4.02)

19. Secondary Outcome: Number of PWD Primary Care Provider Contacts During Study Period
Time Frame: Up to Day 60
Measure: Mean (Standard Deviation); unit: Primary Care Provider Contacts
Arm/Group | QI Program Care | Control
Number analyzed (Participants) | 119 | 96
Primary Care Provider Contacts | 0.64 (0.86) | 0.68 (0.84)

20. Secondary Outcome: Change in Zarit Burden Inventory Score Among Caregivers
Description: 22-item self-assessment of burden experienced by caregivers. Items are ranked on a Likert scale from 0 (never) to 4 (nearly always). The total score is the sum of responses and ranges from 0 to 88, where: 0 - 21 = little or no burden; 21 - 40 = mild to moderate burden; 41 - 60 = moderate to severe burden; and 61 - 88 = severe burden. An increase in scores indicates burden increased during the observational period.
Time Frame: Baseline, Day 60
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | QI Program Care | Control
Number analyzed (Participants) | 117 | 95
score on a scale | 29.65 (16.21) | 26.14 (13.45)

21. Secondary Outcome: Change in Public Health Questionnaire-9 (PHQ-9) Score Among Caregivers
Description: 9-item measurement of depression in which caregivers indicate how often they have been bothered by specific problems over the previous 2 weeks. Items are ranked on 4-point Likert scale ranging from 0 (not at all) to 3 (nearly every day). The total score is the sum of responses and ranges from 0 to 27; higher scores indicate greater severity of depression.
Time Frame: Baseline, Day 60
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | QI Program Care | Control
Number analyzed (Participants) | 119 | 96
score on a scale | 4.8 (5.03) | 4.27 (4.04)

22. Secondary Outcome: Change in Short-Form-12 - Physical Subscale (PCS-12) Score Among Caregivers
Description: 12-item tool that measures functional health and well-being. Two summary scores are reported from the SF-12: a mental component score (MCS-12) and a physical component score (PCS-12). Physical Composite Scores (PCS) are computed using the scores of twelve questions and range from 0 to 100, where a zero score indicates the lowest level of health measured by the scales and 100 indicates the highest level of health.
Time Frame: Baseline, Day 60
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | QI Program Care | Control
Number analyzed (Participants) | 119 | 96
score on a scale | 47.15 (11.13) | 47.13 (11.36)

23. Secondary Outcome: Change in Short-Form-12 - Mental Health Subscale (MCS-12) Score Among Caregivers
Description: 12-item tool that measures functional health and well-being. Two summary scores are reported from the SF-12: a mental component score (MCS-12) and a physical component score (PCS-12). Mental Health Composite Scores (MCS) are computed using the scores of twelve questions and range from 0 to 100, where a zero score indicates the lowest level of health measured by the scales and 100 indicates the highest level of health.
Time Frame: Baseline, Day 60
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | QI Program Care | Control
Number analyzed (Participants) | 119 | 96
score on a scale | 46.63 (11.8) | 47.59 (9.26)

ADVERSE EVENTS:
Time Frame: 60 Days
Description: The Data Safety and Monitoring Board required a focused adverse event (AE) collection process which requires following single AE: a PHQ-9 score worsened by greater than or equal to 5 points during the course of the study. The DSMB required monitoring the following severe AEs: Caregiver attempted suicide; death of caregiver; death of person with dementia a; medical event that may jeopardize the subject, including hospitalization of either the person with dementia or caregiver, suicidal ideation.
Arm/Group | QI Program Care - PWD | QI Program Care - Caregiver | Control - PWD | Control - Caregiver
All-Cause Mortality (participants affected / at risk) | 6/119 | 0/119 | 10/96 | 0/96
Serious Adverse Events (participants affected / at risk) | 26/119 | 3/119 | 34/96 | 4/96
Other Adverse Events (participants affected / at risk) | 21/119 | 5/119 | 9/96 | 1/96
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | QI Program Care - PWD (N=119) | QI Program Care - Caregiver (N=119) | Control - PWD (N=96) | Control - Caregiver (N=96)
Hospitalization (General disorders) | 15 | 0 | 19 | 2
Caregiver severe depression (Increase Score on PHQ-9 [Day 60]) (Psychiatric disorders) | 0 | 2 | 0 | 2
Caregiver suicide idealization (Psychiatric disorders) | 0 | 1 | 0 | 0
Death related (General disorders) | 6 | 0 | 10 | 0
Delirium (Psychiatric disorders) | 5 | 0 | 5 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | QI Program Care - PWD (N=119) | QI Program Care - Caregiver (N=119) | Control - PWD (N=96) | Control - Caregiver (N=96)
Increase in symptoms of dementia (Nervous system disorders) | 7 | 0 | 1 | 0
Change in pre-existing condition (General disorders) | 1 | 4 | 0 | 0
New Diagnosis (General disorders) | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 9 | 0 | 6 | 0
Depressive Symptoms (Score on PHQ-9) (Psychiatric disorders) | 0 | 1 | 0 | 1
Injury not life threatening (Injury, poisoning and procedural complications) | 2 | 0 | 1 | 0
Delirium False Positive (Psychiatric disorders) | 2 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-27): https://cdn.clinicaltrials.gov/large-docs/67/NCT03255967/Prot_SAP_000.pdf